CLINICAL TRIAL: NCT00446160
Title: Proposal for Retrospective Review of an Adult Congenital Heart Surgery Program
Brief Title: Adult Congenital Heart Disease Surgery
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Subhadra Shashidharan, Assistant Professor, Emory University
Other Study IDs: IRB00002790
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Congenital Disorders
Keywords: Congenital Heart Disease; Surgery; Adult
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is now estimated that the number of adults with congenital heart disease in the U.S is over 800,000. Unfortunately, these patients, in some way, have become a lost population. They have congenital abnormalities familiar to a children's hospital, yet have surpassed the age cutoff for admission.

Recently, we have developed a specialized program to care for this unique patient population. Dedicated programs such as ours hope to optimize patient care, consolidate specialized resources, provide sufficient patient numbers for training and maintain expertise and facilitate research in this unique population.

DETAILED DESCRIPTION:
In the United States, approximately 30,000 children are born with congenital heart disease every year. As technology, operative technique, and critical care medicine have improved significantly over the years, more of these children are surviving into adulthood.

Care of the congenital cardiac surgical patient requires a concerted effort on the part of the surgeons, perfusionists, anesthesiologists, intensivists, nurses, respiratory therapists, rehabilitation services and social workers. It is hoped that the same excellent care received in a children's congenital heart surgery program can be continued as these patients graduate into an adult program.

This is a retrospective chart review examining patients over the age of 18 years who have undergone operations for congenital heart disease. The primary interest of the study is to look at the breakdown of our adult congenital program in regards to location, personnel, and case type. All charts reviewed will be of patients who had their surgery at Children's Healthcare of Atlanta or Emory University between January 1, 2000 and December 31, 2006. We will review approximately 225 charts for this study.

The first aim of the study would be to examine the demographics of the adult congenital heart surgery program itself. The following information will be collected:

* Location of the surgery - children's hospital vs adult hospital
* Surgeon - adult cardiac surgeon vs congenital cardiac surgeon

The second aim of the study would be to analyze the types of surgeries being performed. The following information will be collected:

* Pathologic diagnosis
* Number of re-operative sternotomies
* Number of open-heart surgeries

The third aim of the study would be to analyze our outcomes. The following information will be collected:

- Number of surgical mortalities

ELIGIBILITY:
Inclusion Criteria:

* surgery at Children's Healthcare of Atlanta or Emory University between 1.1.2000 and 12.31.2007
* surgery on patients after 18 years to approximately 65 years of age

Exclusion Criteria:

* Those who do not meet inclusion criteria

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective chart review examining patients over the age of 18 years who have undergone operations for congenital heart disease. The primary interest of the study is to look at the breakdown of our adult congenital program in regards to location, personnel, and case type. All charts reviewed will be of patients who had their surgery at Children's Healthcare of Atlanta or Emory University between January 1, 2000 and December 31, 2007. We will review approximately 350 charts for this study.
  Some of the patients have been cared for in the system for many years, first at Egleston and then at Emory. We are only interested in the congenital operations performed on patients after the age of 18 years old up until approximately 65 years of age. Initially these were done at Egleston, although more recently they are being done at Emory.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2000-01; Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
The primary interest of the study is to look at the breakdown of our adult congenital program in regards to location, personnel, and case type. | Retrospective chart review

CONTACTS AND LOCATIONS:
Overall Officials: Subhadra E Shashidharan, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States